CLINICAL TRIAL: NCT02622243
Title: Duration of Bronchoprotection of the Long Acting Muscarinic Antagonists Tiotropium and Glycopyrronium Against Methacholine Induced Bronchoconstriction
Brief Title: Duration of Long Acting Muscarinic Antagonist (LAMA) Bronchoprotection Against Methacholine Challenge
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio REB 15-254
Record Dates: First submitted 2015-11-27; First posted 2015-12-04 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tiotropium (Experimental): 2 inhalations of 2.5mcg/inhalation tiotropium from Respimat inhaler and 1 inhalation of placebo from Breezehaler 1 hour prior to methacholine challenge
  Interventions: Drug: Tiotropium; Device: Respimat; Device: Breezehaler
- glycopyrronium (Experimental): 1 inhalation of 50mcg glycopyrronium from Breezehaler and 2 inhalations from placebo Respimat inhaler 1 hour prior to methacholine challenge
  Interventions: Drug: glycopyrronium; Device: Respimat; Device: Breezehaler

INTERVENTIONS:
Drug: Tiotropium — long acting muscarinic antagonist
  Other Names: Spiriva
  Arms: tiotropium
Drug: glycopyrronium — long acting muscarinic antagonist
  Other Names: Seebri
  Arms: glycopyrronium
Device: Respimat — inhaler device used to deliver active tiotropium or placebo
Device: Breezehaler — inhaler device used to deliver active glycopyrronium or placebo

SUMMARY:
The study will assess the duration of protection of single doses of 2 different long acting muscarinic antagonists against methacholine induced bronchoconstriction.

ELIGIBILITY:
Inclusion Criteria:

* male or female asthmatics > 19 years of age
* baseline methacholine PC20 less than or equal to 4mg/ml
* baseline lung function >65% predicted
* non-smoker and less than 10 pack year smoking history

Exclusion Criteria:

* use of anticholinergic within 30 days of Visit 1
* poorly controlled asthma
* pregnant or nursing
* respiratory illness within 4 weeks of Visit 1
* exposure to an agent that triggered asthma worsening (e.g. allergen) within 4 weeks of Visit 1

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline methacholine bronchoprotection at 96 hours | pre treatment versus 96 hour post treatment
  assessed by dose shift of geometric mean methacholine PC20 data

SECONDARY OUTCOMES:
Change from baseline methacholine bronchoprotection at 1 hour | pre treatment versus 1 hour post treatment
  assessed by dose shift of geometric mean methacholine PC20 data
Change from baseline methacholine bronchoprotection at 24 hours | pre treatment versus 24 hours post treatment
  assessed by dose shift of geometric mean methacholine PC20 data
Change from baseline methacholine bronchoprotection at 48 hours | pre treatment versus 48 hours post treatment
  assessed by dose shift of geometric mean methacholine PC20 data
Change from baseline methacholine bronchoprotection at 72 hours | pre treatment versus 72 hours post treatment
  assessed by dose shift of geometric mean methacholine PC20 data

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
journal publication

REFERENCES:
- [Derived] Blais CM, Davis BE, Cockcroft DW. Duration of bronchoprotection of the long-acting muscarinic antagonists tiotropium & glycopyrronium against methacholine-induced bronchoconstriction in mild asthmatics. Respir Med. 2016 Sep;118:96-101. doi: 10.1016/j.rmed.2016.07.017. Epub 2016 Jul 30. PMID 27578477